CLINICAL TRIAL: NCT04722549
Title: Effects of Butyrate on Affective Processes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Kristin Verbeke, Prof. Dr. Kristin Verbeke, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: S60501- Exp 2
Record Dates: First submitted 2021-01-21; First posted 2021-01-25 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Emotions; Stress; Fear
MeSH Terms: interventions — Butyrates

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants, investigators, and personnel involved in data analyses are blinded to the intervention. Unblinding occurs after all data has been collected AND analysed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo (cellulose)
  Interventions: Dietary Supplement: Placebo
- Butyrate (Active Comparator): Sodium butyrate
  Interventions: Dietary Supplement: Butyrate

INTERVENTIONS:
Dietary Supplement: Placebo — Cellulose
  Arms: Placebo
Dietary Supplement: Butyrate — Sodium butyrate
  Arms: Butyrate

SUMMARY:
The effects of butyrate on psychobiological processes are examined in a sample of healthy volunteers.

DETAILED DESCRIPTION:
The study is an interventional triple-blind, placebo-controlled, parallel group design with 2 arms (placebo, butyrate). Healthy male participants adhere to a low-fiber diet for the duration of the study (11 days). At the baseline study visit, measurements are taken in the lab, including biological samples and psychophysiological measurements. Participants then consume placebo or butyrate for 1 week and revisit the lab on day 11 for a second measurement of the outcomes of interest. Specifically, we investigate the effect of colonic butyrate administration on affective processing, including stress sensitivity and fear-related processes (e.g. extinction learning). Volunteers also respond to questionnaires in relation to mood and GI symptoms, and provide biological samples (saliva, blood, and faecal samples) for analysis of cortisol levels, circulating short chain fatty acids and serum BDNF, and faecal SCFA, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Male participants
* Age range 20-40 years
* BMI range 18.5-25
* Dutch or English as native-language

Exclusion Criteria:

* previous or current neurological, psychiatric, gastrointestinal or endocrine disorders, or other relevant medical history
* current or recent regular medication use
* previous or current substance/alcohol dependence or abuse (> 2 units per day/14 units per week)
* one or more diagnoses based on the mini-international neuropsychiatric interview
* smoking
* night-shift work
* adherence to vegan or vegetarian diets
* use of pre- or probiotics within one month preceding the study
* use of antibiotics within 3 months preceding the study
* previous experience with one of the tasks used in the study

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2022-12-11 (Actual); Study Completion 2022-12-11 (Actual)

PRIMARY OUTCOMES:
Stress sensitivity (cortisol) | through study completion, on average 1 year and 5 months
  Induction of cognitive, physical, and social stress using Maastricht Acute Stress Test. Stress hormone cortisol is quantified by gathering multiple saliva samples throughout the stress induction and recovery during both pre-intervention and post-intervention visit.

SECONDARY OUTCOMES:
Stress sensitivity (subjective) | through study completion, on average 1 year and 5 months
  Induction of cognitive, physical, and social stress using Maastricht Acute Stress Test. Participant rate how much stress, discomfort, and pain they feel on a 10-cm visual analogue scale, with higher values indicating greater stress, discomfort, and pain. This is done prior to stress induction, in the middle, and at the end at both pre- and post-intervention visits.
Cortisol awakening response | through study completion, on average 1 year and 5 months
  Measuring chronic stress by quantifying cortisol in morning samples (5 samples taken form the moment of waking every 15 minutes for 1 hour) on the morning of the pre- and post-intervention visits.
Fear | through study completion, on average 1 year and 5 months
  Exploring fear-related processes (conditioning, extinction, recall, and renewal) by means of a computerised task. Fear response is measured using skin conductance, and a skin conductance response is calculated.
Fear (subjective) | through study completion, on average 1 year and 5 months
  Exploring fear-related processes (conditioning, extinction, recall, and renewal) by means of a computerised task. Fear response is measured subjectively by asking participants to indicate their expectancy of an aversive stimulus.
Positive and Negative Affect Schedule (PANAS) | through study completion, on average 1 year and 5 months
  Assessing ratings on the subscales of PANAS, positive and negative affect. PA subscale scores range between 10-50, with higher scores indicating better outcome.
  NA subscale scores range between 10-50, with higher scores indicating worse outcome.
Perceived Stress Scale (PSS) | through study completion, on average 1 year and 5 months
  Assessing ratings on PSS. Scores range between 0-40 with higher scores indicating worse outcome.
Depression, anxiety, and stress scales (DASS-21) | through study completion, on average 1 year and 5 months
  Assessing ratings on the subscales of DASS-21, depression, anxiety, and stress subscales.
  Higher scores on these subscales indicates a worse outcome.
  Normal (depression: 0 - 4; anxiety: 0 - 3; stress: 0 - 7), Mild (depression: 5 - 6; axiety: 4 - 5; stress: 8 - 9), Moderate (depression: 7 - 10; anxiety: 6 - 7; stress: 10 - 12), Severe (depression: 11 - 13; anxiety: 8 - 9; stress: 13 - 16), Extremely Severe (depression: 14 +; anxiety: 10 +; stress: 17 +).
Leiden Index of Depression Sensitivity-Revised (LEIDS-R) | through study completion, on average 1 year and 5 months
  Assessing ratings on the subscales of LEIDS-R and its total score. This is a self-report on cognitive reactivity comprised of 34 items with six subscales. Hopelessness/suicidality; Acceptance/Coping; Aggression; Control/Perfectionism; Risk Aversion; Rumination.
Gastrointestinal symptom rating scale (GSRS) | through study completion, on average 1 year and 5 months
  Assessing ratings on the subscales of GSRS and its total score. It has 5 subscales (Reflux, Diarrhea, Constipation, Abdominal Pain, and Indigestion Syndrome). Subscale scores range from 1 to 7 and higher scores indicates a worse outcome.
Serum SCFA | through study completion, on average 1 year and 5 months
  Quantification of serum SCFA (μM) at pre- and post-intervention
Faecal SCFA | through study completion, on average 1 year and 5 months
  Quantification of faecal SCFA in samples provided at pre- and post-intervention
Serum BDNF | through study completion, on average 1 year and 5 months
  Quantification of fasting serum BDNF levels (µg/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Verbeke, Prof, Principal Investigator — kristin.verbeke@kuleuven.be
Locations (1):
- UZ Leuven/Stresslab, Leuven, I Am Not in the U.S. Or Canada, Belgium

IPD SHARING:
Plan to Share IPD: Undecided